CLINICAL TRIAL: NCT05787028
Title: Safety, Tolerability and Pharmacokinetics of AD16 Tablets in Adult Healthy Subjects After Single Administration
Acronym: AD16
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: South China Center For Innovative Pharmaceuticals (Other)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCCIP-AD16-2018-01
Record Dates: First submitted 2023-03-01; First posted 2023-03-28 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: A single-center, randomized, placebo-controlled, double-blind, dose-increasing study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AD16 (Experimental): The experimental group received AD16, which was a tablet with a dosage form of 10mg/tablet. Take warm water orally on an empty stomach in the morning, once a day.7 dosing cohorts will receive a single oral dose of AD16.
  Interventions: Drug: AD16 5mg、10mg、20mg、30mg、40mg、60mg、80mg
- placebo (Placebo Comparator): The placebo group received AD16 placebo, which was a tablet with a dosage form of 10mg/tablet. Take warm water orally on an empty stomach in the morning, once a day.
  7 dosing cohorts will receive a single oral dose of AD16 placebo.
  Interventions: Drug: AD16 placebo 5mg、10mg、20mg、30mg、40mg、60mg、80mg

INTERVENTIONS:
Drug: AD16 5mg、10mg、20mg、30mg、40mg、60mg、80mg — Take one AD16 tablet in the morning
  Arms: AD16
Drug: AD16 placebo 5mg、10mg、20mg、30mg、40mg、60mg、80mg — Participants will take a placebo pill matching AD16 once in the morning
  Arms: placebo

SUMMARY:
The primary objective of this study was to evaluate the safety, tolerability and pharmacokinetic characteristics of single administration of AD16 tablets in healthy adults under fasting conditions, and the secondary objective was to preliminarily evaluate the material balance of single administration of AD16 tablets in fasting conditions.

The study is divided into two parts: preliminary test and formal test. The formal trial was a single-center, randomized, placebo-controlled, double-blind, dose-increasing study, with 5 dose groups (5mg, 10mg, 20mg, 30mg and 40mg, respectively).

Ten subjects (male and female) were enrolled in each dose group, of which 8 received the experimental drug and 2 received placebo.

Urine and fecal samples were collected in the 20mg dose group for material balance study.Urine and fecal samples were collected in the 20mg dose group for material balance study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects were aged 18-45 years (including boundary values), male and female.
2. Weight ≥50kg (male) or ≥45kg (female), and body mass index (BMI) of 19-24kg/m2 (including the boundary values at both ends).
3. Have fully understood this study, voluntarily participated in it, and signed the Informed Consent.
4. Subjects are able to communicate well with researchers and complete the study according to protocol.
5. The subjects were deemed to be in good health based on physical examination, medical history, vital signs, electrocardiogram, chest X-ray, abdominal ultrasound, and laboratory tests.
6. Subject (including partner) is willing to have no pregnancy plan for the next 30 days (female subject) or 90 days (male subject) and is willing to use effective contraception.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen, hepatitis C antibody, syphilis antibody or HIV antibody.
2. The patient has symptoms or related history of any serious disease, including but not limited to heart, liver, kidney, or other acute or chronic digestive tract or respiratory tract diseases, as well as diseases of the blood, endocrine, neurological, psychiatric and other systems, or any other disease or physiological condition that can interfere with the study results.
3. A history of postural hypotension with frequent episodes.
4. A history of frequent nausea or vomiting due to any cause.
5. Any clear history of drug or food allergies, especially allergies to ingredients similar to the drugs in this study.
6. Have special dietary requirements and cannot comply with the uniform diet provided by the clinical research center.
7. Previous drug abuse history or positive urine drug screening during screening period.
8. Smokers who smoked more than 5 cigarettes a day in the 3 months before the test.
9. Heavy drinkers or regular drinkers in the 6 months prior to the study screening, who drank more than 14 units of alcohol per week (1 unit of alcohol ≈360 mL beer or 45 mL 40% spirits or 150 mL wine) or had a positive alcohol breath test during the screening period.
10. Excessive consumption of tea, coffee (more than 6 cups) and/or caffeinated beverages (more than 1L) per day.
11. Surgical procedures, transfusions of blood or blood components in the month prior to study screening.
12. Blood loss or donation of more than 400 mL in the 2 months prior to screening.
13. Participated in other clinical studies and took experimental drugs within 3 months prior to study screening.
14. Study participants who had received any medication in the 28 days prior to screening.
15. Pregnant or lactating women or women who have had unprotected sex within 14 days.
16. Those unable to complete the study for other reasons or deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | day-7 to day3
  The number of adverse events
Serious adverse events | day-7 to day3
  The number of serious adverse events
Number of participants with abnormal laboratory test results | Screening period (day-7 to day-2) and day3
  Laboratory tests include Blood routine, blood biochemistry, coagulation function and urine routine
Number of participants with abnormal vital signs | day-7 to day3
  Pulse, blood pressure, body temperature and respiratory rate were observed at different time points before and after medication.
Number of participants with abnormal 12-lead electrocardiogram readings | Screening period (day-7 to day-2) and day3
  abnormal 12-lead electrocardiogram readings
Number of participants with abnormal physical examination findings | Screening period (day-7 to day-2) and day3
  The skin, mucosa, lymph nodes, head, neck, chest, abdomen, spine/limbs and nervous system were observed at different time points before and after medication.
Concomitant Medication | up to day3
  Any concomitant medication
Tmax of AD16 | day1 to day3
  Time to reach the maximum (peak) plasma concentration following drug administration
Cmax of AD16 | day1 to day3
  Maximum (peak) plasma drug concentration
t1/2z of AD16 | day1 to day3
  Elimination half-life (to be used in a one-compartment or noncompartmental model)
AUC 0-∞ of AD16 | day1 to day3
  AUC 0-∞ is defined as the concentration of drug extrapolated to infinite time (area under the plasma concentration versus time curve extrapolated to infinite time).
  area under curve(AUC)
AUC 0-t of AD16 | day1 to day3
  AUC 0-t is defined as the concentration of drug from time zero to the last quantifiable concentration.area under curve(AUC)
CL/F of AD16 | day1 to day3
  CL/F is defined as the ratio of total clearance(CL) to bioavailability(F).
  administration
Vd/F of AD16 | day1 to day3
  Apparent volume of distribution after non-intravenous administration
λz of AD16 | day1 to day3
  Terminal disposition rate constant/terminal rate constant
Mean retention time（MRT ）of AD16 | day1 to day3
  Mean retention time from first dosing to t hours or mean retention time from first dosing to infinity

SECONDARY OUTCOMES:
Ae | day-3 to day3
  The amount of drug excreted in urine at t hours after administration The amount of drug excreted by fecal sample at t hours after administration
Fe0-t | day-3 to day3
  Cumulative excretion rate of drugs through urine Cumulative rate of drug excretion through feces
Renal clearance | day-3 to day3
  Renal clearance of drug from plasma

CONTACTS AND LOCATIONS:
Locations (1):
- The Central South University Xiang Ya Hospital, Changsha, China

REFERENCES:
- [Derived] Peng D, Xu S, Zou T, Wang Y, Ouyang W, Zhang Y, Dong C, Li D, Guo J, Shen Q, Hu X, Zhou W, Li X, Qin Q. Safety, tolerability, pharmacokinetics and effects of diet on AD16, a novel neuroinflammatory inhibitor for Alzheimer's disease: a randomized phase 1 study. BMC Med. 2023 Nov 23;21(1):459. doi: 10.1186/s12916-023-03126-9. PMID 37996817